CLINICAL TRIAL: NCT01925846
Title: Association of Type Three Secretion System (T3SS) of Pseudomonas Aeruginosa With Pathogenesis of Contact Lens-Associated Microbial Keratitis (CLMK)
Brief Title: Pseudomonal Type Three Secretion System and Contact Lens Associated Microbial Keratitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201212003RINC
Record Dates: First submitted 2013-08-16; First posted 2013-08-20 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Keratitis; Infectious Disease (Manifestation)
Keywords: Pseudomonas aeruginosa; type three secretory system; contact lens associated microbial keratitis
MeSH Terms: conditions — Keratitis; Communicable Diseases; Pseudomonas Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Microbial infection of the cornea, also known as microbial keratitis, causes severe corneal inflammation that could result in permanent visual loss. Contact lens wear is the strongest risk factor related to microbial keratitis in developed countries. The most commonly isolated pathogen of contact lens associated microbial keratitis (CLMK) is Pseudomonas aeruginosa, which accounts for over one third of the cases. Among the various virulence factors involved in the pathogenesis of pseudomonal keratitis, a secretion system known as type three secretion system (T3SS) secretes toxins that damage the host cells. ExoS is a bifunctional exotoxin with GTPase-activating protein (GAP) activity and ADP ribosyl transferase (ADPRT) activity. It results in an invasive phenotype of P. aeruginosa causing a relatively slower host cell death with intracellular invasion and possibly proliferation of bacterium. In contrast, ExoU expressing strains carries a cytotoxic phenotype that causes rapid host cell lysis due to its phospholipase activity. Previously, cytotoxic strains were reported to be more commonly found in patients with pseudomonal keratitis and were highly correlated with multidrug resistance.

In order to understand the pathogenesis of CLMK, especially pseudomonal related CLMK, we proposed to recruit 180 volunteers who will wear different contact lens materials. We then collect the used contact lens and analyze 1) the microbiota on the used contact lens; 2) the bacterial-contact lens adhesion of wild strains, pscC mutant strains (T3SS needle-comples mutant), cytotoxic strain, and invasive strain P. aeruginosa; 3) the effect of shearing forces on bacterial-contact lens adhesion; 4) the bacteriocidal effect of multipurpose solution on different strains of P. aeruginosa.

DETAILED DESCRIPTION:
Subject recruitment

The inclusion criteria includes:

1. age 20-35 years old
2. myopia less than -6.00D and astigmatism less than -1.50D
3. previous soft contact lens wear discontinued for at least 2 weeks.

Exclusion criteria includes:

1. subjects with previous RGP wear
2. any ocular inflammation or infection, proved dry eye syndrome, glaucoma, ocular trauma or surgery, and topical medication instillation
3. diabetic mellitus
4. pregnancy
5. status post corneal refractive surgery

The aim and purpose of this study will be thoroughly explained to the potential participants. Informed consent will be obtained from all enrolled subjects. This study will be approved by our Institutional Review Board and adheres to the tenets of the Declaration of the Helsinki. A minimal of 12 subjects per group is required to show a difference in the microbiota for one classification level or more at a significance level of 0.05 and a power of 90%. Thus, the goal is to recruit 15 volunteers to wear each type of contact lens and 180 subjects totally for this study.

The recruitment will be divided into three stages. At the first stage, we will test 4 types of silicone hydrogel contact lenses, followed by testing 5 types of color-tinted hydrogel lenses at the second stage and 3 types of hydrogel lenses at the third stage. (T = types of lenses, which equals 4,5 and 3 at stage one, two and three).

At each stage, we will recruit subjects to certain amount (M) each time (M＝N×T , N equals 1,2,3…to 15). M subjects will then be randomized, equally distributed to wear T types of lenses by the random number method. Until the required case numberis achieved at the first stage, we will proceed to the second and the third stage with the same stratified randomization methods.( required case number, ΣM, equals 60, 75 and 45 at stage one, two and three).

Subjects are fitted with the soft contact lenses and are expected to wear the lenses for at least 6-8 hour per day. Standardized hand hygiene and lens care regimen are thoroughly explained to each subject to insert the contact lens. Each subject enrolled will be provided with the soft contact lenses without charge. After wear each day, the contact lenses must be returned and collected for material analysis.

ELIGIBILITY:
Inclusion Criteria:

1. age 20-35 years old
2. myopia less than -6.00D and astigmatism less than -1.50D
3. previous soft contact lens wear discontinued for at least 2 weeks. -

Exclusion Criteria:

1. subjects with previous RGP wear
2. any ocular inflammation or infection, proved dry eye syndrome, glaucoma, ocular trauma or surgery, and topical medication instillation
3. diabetic mellitus
4. pregnancy
5. status post corneal refractive surgery -

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In order to understand the pathogenesis of CLMK, especially pseudomonal related CLMK, we proposed to recruit 180 volunteers who will wear different contact lens materials. We then collect the used contact lens and analyze 1) the microbiota on the used contact lens; 2) the bacterial-contact lens adhesion of wild strains, pscC mutant strains (T3SS needle-comples mutant), cytotoxic strain, and invasive strain P. aeruginosa; 3) the effect of shearing forces on bacterial-contact lens adhesion; 4) the bacteriocidal effect of multipurpose solution on different strains of P. aeruginosa.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
bacterial adhesion assay | after co-culture for two hours

SECONDARY OUTCOMES:
Identification of bacterial colonization to worn contact lenses | after the CL been worn for 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: HU FR Hu, professor, Study Chair
Locations (1):
- Department of Ophthlamology, National Taiwan University Hospital, Taipei, Taiwan